CLINICAL TRIAL: NCT00451308
Title: Induction of Labor With a Foley Catheter Balloon: A Randomized Trial Comparing Inflation With 30ml and 60ml
Brief Title: Induction of Labor With a Foley Balloon Catheter: Inflation With 30ml Compared to 60ml
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H4114729401-01
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Induction of Labor
Keywords: Induction of labor; vaginal delivery; cesarean section; foley balloon cathether; method of labor induction; perinatal outcomes
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Foley balloon wih 60cc fluid
  Interventions: Procedure: Induction of labor with foley balloon - 60cc of saline
- 2 (Active Comparator): Foley balloon with 30cc
  Interventions: Procedure: Induction of labor with foley balloon with 30cc

INTERVENTIONS:
Procedure: Induction of labor with foley balloon - 60cc of saline — 60 cc of fluid
  Arms: 1
Procedure: Induction of labor with foley balloon with 30cc — 30cc of saline in foley
  Arms: 2

SUMMARY:
The rate of labor induction is rising throughout the United States for a variety of reasons. Medical conditions that lead to increased risk of prolonging the pregnancy to both mother and fetus are not infrequent. In addition, elective deliveries are becoming more common. Foley balloon catheter placement is a common method used for labor induction in women with an unfavorable cervical assessment. There are several studies using various volumes of Foley balloon catheters for labor induction ranging from 30ml to 80ml, however, there are no studies replicating the findings of the largest study comparing 2 different volumes in the balloon. The investigators plan to compare instillation of 30ml of sterile saline versus 60ml in a Foley balloon catheter for women undergoing induction of labor with an unfavorable cervix. The investigators will observe the following outcomes: rate of delivery within 24 hours, cervical dilation after foley balloon catheter expulsion, insertion to balloon expulsion interval, induction to delivery time interval, peak oxytocin requirement, presence of infection or meconium, cesarean delivery rate, operative vaginal delivery rate, indication for operative vaginal or cesarean delivery, cervical laceration rate, placental abruption rate, 5-minute Apgar score, and umbilical cord arterial blood pH and base excess.

DETAILED DESCRIPTION:
All potential candidates will be approached for the study and undergo written consent if willing to participate. Each candidate will be randomized to 30ml or 60 ml Foley balloon catheter volume. A random number generator will be used and within a sealed envelope will be placed the assignment. Nulliparous and multiparous patients will be randomized separately. The patient will be positioned for a standard cervical exam - either for digital or speculum exam, depending on the individual patient preference and provider choice. For digital exam, a sterile Foley balloon catheter will be digitally placed in the endocervical canal, into the extraamniotic space (between the fetal head, external to the unruptured amniotic sac, above the internal os of the cervix). For speculum exam, the cervix is wiped three times with a Betadine cleansing solution, and a sterile Foley balloon catheter bulb will be placed under direct visualization into the endocervical canal, into the extraamniotic space. Once the balloon is in place the provider inserts 30ml of sterile saline. The provider then leaves the room. The patient's nurse opens the envelope and if the patient is allocated to the 60ml volume group, the nurse adds an additional 30ml of sterile saline. If the patient is in the 30ml group, the RN staff will simulate placement of additional saline into the foley balloon without actually placing any additional saline in order to also blind the patients to their assigned group. The MD/CNM providers will then return to the room, blinded to the inflation of the Foley balloon, and the balloon catheter will be placed under tension by taping the external end to the patient's inner thigh. Oxytocin will be started within 30 minutes of the Foley balloon catheter placement, using the standard intravenous oxytocin protocol. Additional manual traction on the Foley balloon catheter will be performed every 30 minutes until Foley balloon catheter expulsion. A sterile cervical exam will be performed after spontaneous Foley catheter expulsion to evaluate post-balloon cervical dilation. No further procedures or tests specific to this study will be required beyond this point; only data collection on the above study outcomes during the remaining course of the patient's labor will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women, pregnant, term gestation (>37 weeks), undergoing induction of labor, cervical exam acceptable as a candidate for Foley balloon catheter placement (Bishop score <5), cephalic fetal presentation.

Exclusion Criteria:

* Regular contractions on admission, rupture of membranes, previous uterine scar, low-lying placenta (measured <3cm to internal os), Bishop score > 5, contraindication to attempt at vaginal birth, non-English/Spanish speaking, unable to give consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2006-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Rate of vaginal delivery within 24 hours | within 24 hours

SECONDARY OUTCOMES:
Cervical dilation after Foley balloon catheter expulsion | within 24hours
Time to catheter expulsion | hours
Duration of the first stage of labor | hours
Time interval from induction to active labor | hours
Induction to delivery interval | hours
Presence of abnormal vaginal bleeding | hours
Peak oxytocin requirement during induction and labor augmentation | hours
Epidural utilization, diagnosis of chorioamnionitis | hours
Meconium stained amniotic fluid, placental abruption | hours
Cesarean delivery rate, operative vaginal delivery rate | hours
Indication for operative vaginal or cesarean delivery | hours
Rate of cervical laceration | hours
Birthweight | hours
5 minute Apgar score | hours
Umbilical cord arterial blood pH analysis | hours

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Caughey, MD,PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Department of Obstetrics, Gynecology and Reproductive Sciences, San Francisco, California, United States

REFERENCES:
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Delaney S, Shaffer BL, Cheng YW, Vargas J, Sparks TN, Paul K, Caughey AB. Labor induction with a Foley balloon inflated to 30 mL compared with 60 mL: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1239-1245. doi: 10.1097/AOG.0b013e3181dec6d0. PMID 20502296